CLINICAL TRIAL: NCT06232486
Title: Association Between Serum Vitamin D and Postherpetic Neuralgia, A Prospective Observation Study.
Brief Title: Relationship Between Serum Vitamin D Levels and Postherpetic Neuralgia.
Status: Active, not recruiting | Type: Observational
Sponsor: Feng Gao (Other)
Responsible Party: Sponsor-Investigator, Feng Gao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20231251
Record Dates: First submitted 2023-12-25; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Postherpetic Neuralgia
Keywords: Herpes zoster,post-herpes zoster,Vitamin D,
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Herpes zoster patients: The patient was diagnosed with herpetic neuralgia and the course of disease was ≤3 months;

SUMMARY:
1. The correlations of serum vitamin D level, serum calcium level and osteoporosis degree with disease severity, treatment response, incidence of Post-Herpes zoster(PHN) and disease prognosis in Herpes zoster(HZ) patients were studied.
2. To investigate the role of inflammation-related factors and immune-related factors in the occurrence and development of HZ mediated by low vitamin D level.

DETAILED DESCRIPTION:
Herpes zoster is a neuropathic disease which induce by the varicella-herpes virus reactivation.and postherpetic neuralgia (PHN) is the most common complication. Currently,the mechanism of herpes zoster still unclearly even though there had much study about it .Vitamin D is an essential vitamin for human body, which has the function of maintaining calcium and phosphorus homeostasis and immune regulation. Vitamin D is a natural antiviral substance, and vitamin D deficiency can affect the body's antiviral ability, thereby promoting varicella-zoster virus(VZV) reactivation, and may promote the development of PHN through continuous neuroinflammation. Therefore, vitamin D level may be related to the occurrence and progression of HZ. this study intends to use an observational cohort study design to investigate the correlation of serum vitamin D level and osteoporosis degree with the severity of the herpes zoster disease, Although we plan to further explore the role of inflammatory state in this process.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* The patient was diagnosed with herpetic neuralgia and the course of disease was ≤3 months.
* Can cooperate with the completion of inquiry and scale evaluation.

Exclusion Criteria:

* Severe spinal disease (fracture, malignancy, acute or chronic infection) confirmed by previous spinal surgery or imaging.
* Previous history of head trauma.
* Have autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis, leucothrombocytopenia).
* Suffering from mental disorders, intellectual disability, epilepsy and other diseases.
* A history of substance abuse, drug abuse or alcohol abuse.
* Pregnant or breastfeeding women.
* And recent participation in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with herpes zoster who were hospitalized in the Department of Pain Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology from October 2023 to October 2025 were selected.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D levels | herpetic neuralgia <3 month
  Vitamin D deficiency: < 20 nmol/L. Vitamin D deficiency: 20-30 nmol/L. Normal vitamin D: > 30 nmol/L.

SECONDARY OUTCOMES:
C-reactive protein | Day 2 in the hospital
  An according to early infection stricture in serum.When CRP>20mg/l is considered abnormally level .
Lymphocytes | Day 2 in the hospital
  Lymphocytes is considered an label of virus infection when it outlier.
Red blood cell distribution width,RDM(fl) | Day 2 in the hospital
  It is a reflects the inhomogeneity of red cell size.
Red blood cell count,RBC | Day 2 in the hospital
  One of main recording to diagnosis of anemia . nomal mal (4-5.5)×10-12/L. nomal femal (3.5-5.0)×10-12/L.
Mean red cell volum,MVC | Day 2 in the hospital
  It is a label of red cell size.normal range from 80 to 100fl.
Creatinine | Day 2 in the hospital
  It is a metabolite of muscle and there are have many reasons induce creatinine rise,such as chronic or acute kidney damage,Medicine side effect.normal range:53-106umol/l.
Albumin | Day 2 in the hospital
  It is a protein that is found in many animal tissues and serum.The normal range 35-50g/L.
Alkaline phosphatase | Day 2 in the hospital
  Alkaline phosphatase (ALP or AKP) is an enzyme that is widely distributed in human liver, bone, intestine, kidney, placenta and other tissues and is excreted from the liver to the bile.normal male: 45~125U/L；normal female:20~49岁35~100U/L
Uric acid | Day 2 in the hospital
  Uric acid is the end product of purine metabolism. It is a trioxa purine, and its alcohol form is weakly acidic.normal male:150～416μmol/L，normal female:89～357μmolL
Blood glucose | Day 2 in the hospital
  The production and utilization of blood sugar in normal people are in a state of dynamic balance, maintaining a relatively stable level, which is because the source and route of blood sugar are roughly the same result.Fasting blood-glucose(FBG):4.4~6.1mmol/L。
diastolic blood pressure, | Day 2 in the hospital
  An indicator in blood pressure measurement that indicates the pressure of the heart's arterial blood against the vessel walls during diastole. It is usually measured in millimeters of mercury (mmHg).
systolic blood pressure | Day 2 in the hospital
  A type of blood pressure that refers to the pressure of blood against the artery walls when the heart contracts. It is often used as a measure of cardiovascular health(mmHg).
total cholesterol | Day 2 in the hospital
  The sum of all cholesterol in the blood, including LDL cholesterol and HDL cholesterol. High levels of total cholesterol may increase the risk of cardiovascular disease.normal range：<5.18mmol/L（<200mg/dl）
triglycerides | Day 2 in the hospital
  Triglyceride (TG) is a constituent of lipids, which is formed by glycerol and three fatty acids. normal range<1.70mmol/L.
serum Ca2+ level | Day 2 in the hospital
  Ionic calcium refers to the concentration of calcium ions in the blood, also known as serum calcium. Normal levels of ionic calcium maintain a stable range in the blood, generally 2.1-2.6 mmol/L(or 8.5-10.5 mg/dL).
Cellular immune indexes C3 | Day 2 in the hospital
  Complement C3 can promote phagocytic cells to move to promote phagocytosis, promote B cell proliferation, and have a solubilization effect on soluble immune complex.
Cellular immune indexes C4 | Day 2 in the hospital
  Complement C4 is an important component of the classical activation pathway of complement, which is divided into C4a and C4b. The release of C4a can induce mast cells to release histamine, increase the permeability of blood vessels and cause local exudative inflammation. C4b mainly plays a role in mediating the complement cascade, promoting phagocytosis, participating in preventing the deposition of immune complexes, and neutralizing viruses.
interleukin(IL)-10 | Day 2 in the hospital
  Interleukin-10 is a multi-cellular, multifunctional cytokine that regulates cell growth and differentiation, participates in inflammatory and immune responses, and is a recognized inflammatory and immunosuppressive factor.
interleukinIL-6 | Day 2 in the hospital
  The target cells of IL-6 action are many, including macrophages, hepatocytes, quiescent T cells, activated B cells and plasma cells.
interleukinIL-8 | Day 2 in the hospital
  Interleukin-8, or IL-8 for short, is a cytokine in the family of chemokines. Its role in participating in and regulating the physiological and pathological processes of human reproduction has been confirmed, and one of its mechanisms is to bind to its specific receptors.
tumor necrosis factor(TNF)-a | Day 2 in the hospital
  TNF-α, also known as cachexin and TNFSF1A, is an adipokine involved in systemic inflammation and is one of the cytokines that stimulate the acute phase response. TNF-α transmits information to the nucleus through specific receptors on the cell membrane, thus producing complex biological activities such as promoting cell proliferation and differentiation, immune regulation, inflammation mediation, and anti-tumor.
Bone mineral density T value | Day 2 in the hospital
  Bone mineral density T value,present the bone density to predict osteoporosis.
magnetic resonance imaging | Day 2 in the hospital
  Results of MRI examination,exclude tumor or infection
cluster of differentiation 4(CD4)+ | Day 2 in the hospital
  CD4 cells, refers to the surface of the CD4+T molecule T lymphocytes, is an important immune cell in the human immune system, because the HIV attack object is CD4+T cells, so its detection results on the AIDS treatment effect and the judgment of the patient's immune function has an important role.
cluster of differentiation 8(CD8)+ | Day 2 in the hospital
  CD8+T cells generally refer to cytotoxic T lymphocytes. Cytotoxic T lymphocytes (CTL), a subdivision of white blood cells, are specific T cells that secrete various cytokines to participate in immune function.
numeric rating scale(NRS) | Day 2 in the hospital
  The NRS pain Score is an exponential scale that uses 0 to 10 to represent different levels of pain, 0 being painless and 10 being severe, and asks the patient how bad the pain is, or to circle a number that best represents their pain.
numeric rating scale(NRS) | After the therapy in hospital
  The NRS pain Score is an exponential scale that uses 0 to 10 to represent different levels of pain, 0 being painless and 10 being severe, and asks the patient how bad the pain is, or to circle a number that best represents their pain.
numeric rating scale(NRS) | After the therapy 1 month
  The NRS pain Score is an exponential scale that uses 0 to 10 to represent different levels of pain, 0 being painless and 10 being severe, and asks the patient how bad the pain is, or to circle a number that best represents their pain.
numeric rating scale(NRS) | After the therapy 2 month
  The NRS pain Score is an exponential scale that uses 0 to 10 to represent different levels of pain, 0 being painless and 10 being severe, and asks the patient how bad the pain is, or to circle a number that best represents their pain.
numeric rating scale(NRS) | After the therapy 3 month
  The NRS pain Score is an exponential scale that uses 0 to 10 to represent different levels of pain, 0 being painless and 10 being severe, and asks the patient how bad the pain is, or to circle a number that best represents their pain.
DN4 | Day 2 in the hospital
  A table of pain assesment that mainly about neuropathic pain.
DN4 | After therapy in hospital
  A table of pain assesment that mainly about neuropathic pain.
DN4 | After therapy 1 month
  A table of pain assesment that mainly about neuropathic pain.
DN4 | After therapy 2 month
  A table of pain assesment that mainly about neuropathic pain.
DN4 | After therapy 3 month
  A table of pain assesment that mainly about neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided